CLINICAL TRIAL: NCT05485610
Title: Effect of NMN (Nicotinamide Mononucleotide) Intervention on Patients With Diminished Ovarian Reserve (Including Premature Ovarian Insufficiency)
Brief Title: Effect of NMN (Nicotinamide Mononucleotide) on Diminished Ovarian Reserve (Including Premature Ovarian Insufficiency)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M2022262
Record Dates: First submitted 2022-06-20; First posted 2022-08-03 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-06

CONDITIONS: Diminished Ovarian Reserve; Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMN intervention (Experimental): 3 months of NMN
  Interventions: Dietary Supplement: NMN intervention
- Placebo (Placebo Comparator): 3 months of NMN-free placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NMN intervention — NMN capsules (total of 600mg/day) for 3 months
  Arms: NMN intervention
Other: Placebo — NMN-free placebo capsules for 3 months
  Arms: Placebo

SUMMARY:
The purpose of the study is to understand the effect of nicotinamide mononucleotide (NMN) on patients with diminished ovarian reserve (including premature ovarian insufficiency).

DETAILED DESCRIPTION:
This study aims to evaluate the effects of NMN on reproductive endocrine, immune homeostasis, and reproductive outcomes in women with DOR (including POI), and to explore its underlying mechanisms to provide the intervention strategies for DOR (including POI).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are 20 to 40 years old.
2. The concentrations of anti-Mullerian hormone < 1.1 ng/ml, the values of antral follicle count range from less than 5 to less than 7 and two recordings of serum concentrations of day-3 follicle-stimulating hormone (FSH) ≥10 IU/L.
3. Individuals who can insist on continuous monitoring in the outpatient clinic.
4. Individuals who are not participating in other research projects currently or 3 months before the intervention.

Exclusion Criteria:

1. Individuals who are during pregnant, lactation or menopause.
2. Individuals who had non-46-XX karyotype, or attributed to known genetic etiology.
3. Individuals who had pelvic surgery.
4. Cancer patients or receiving chemo/radiotherapy treatment within the past 5 years.
5. Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
6. Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.
7. Use of medications or traditional Chinese medicine that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 3 months.
8. Individuals who take niacin, nicotinamide, or other vitamin B3-related supplementation, or other supplementation such as coenzyme Q10, vitamin E currently or within the past 3 months.
9. Use of antibiotics, probiotics, or prebiotics that affect the flora within the past 3 months.
10. Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.
11. A medical history of severe cardiovascular and cerebrovascular diseases.
12. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.
13. Individuals who drink more than 15g of alcohol per day or have a smoking habit.
14. Individuals who need drug treatment for any mental illness such as epilepsy and depression.
15. Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.
16. Unable or unwilling to follow the study protocol.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The comparison of the gut microbiota composition | before and after 2, 8, 12 weeks of intervention
  Determination the gut microbiota composition change of stool samples between placebo group and intervention group by 16S metagenomic.
The alterations of gut metabolites | before and after 2, 8, 12 weeks of intervention
  Determination the alterations of gut metabolites before and after NMN intervention by metabolomics.
Blood sugar level | before and after 2, 8, 12 weeks of intervention
  Changes in plasma glucose concentration after the intervention.
Fasting insulin | before and after 2, 8, 12 weeks of intervention
  Changes in plasma insulin concentration after the intervention.
Endocrine hormones including AMH | before and after 3 months of intervention
  Changes in endocrine hormones including AMH levels in serum after the intervention.
Ovarian volume | before and after 3 months of intervention
  The size of each ovary will be determined using transvaginal ultrasonography for each participant in early follicular phase.
Follicle number | before and after 3 months of intervention
  The number of all antral follicles in each ovary will be determined using transvaginal ultrasonography for each participant.
Blood NAD+ level | before and after 2, 8, 12 weeks of intervention
  Changes in whole blood NAD+ level after the intervention.
Changes in NAD-related metabolites in urine | before and after 2, 8, 12 weeks of intervention
  Determination the changes of NAD-related metabolites in urine before and after NMN intervention by metabolomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Patients' information is requested to be confidential.